CLINICAL TRIAL: NCT03003442
Title: Investigation of the Acute and Chronic Effects of Supradyn® Energy 3RDA on Ratings of 'Fatigue/Stress', Substrate Metabolism and Blood Biomarkers of Recovery, as a Consequence of Exercise and Metabolically Demanding Cognitive Tasks
Brief Title: Effects of Supradyn® Energy 3RDA on Fatigue/Stress, Substrate Metabolism During Exercise and Demanding Cognitive Tasks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 18769
Record Dates: First submitted 2016-11-22; First posted 2016-12-28 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: Multivitamin/mineral; Exercise; Fatigue; Stress; Arousal; Energy expenditure; Recovery biomarkers; Cognition
MeSH Terms: conditions — Calcinosis; Motor Activity; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supradyn® Energy 3RDA (Experimental): Supradyn® Energy 3RDA, 1 multivitamin/mineral tablet administered by mouth daily for 28 days
  Interventions: Dietary Supplement: Supradyn® Energy 3RDA
- Placebo (Placebo Comparator): Placebo, 1 tablet administered by mouth daily for 28 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Supradyn® Energy 3RDA — Multivitamin/mineral containing co-Q10
  Arms: Supradyn® Energy 3RDA
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Investigation of the acute and chronic effects of Supradyn® Energy 3RDA on subjective ratings of 'fatigue/stress', substrate metabolism and blood biomarkers of recovery, as a consequence of exercise and metabolically demanding cognitive tasks.

DETAILED DESCRIPTION:
Supplementation with vitamins and minerals has been shown to enhance energy production, metabolism, and mood state. It is thought that they may also aid recovery from challenging physical and psychological tasks following both acute and chronic supplementation. The present study will investigate the effects of a multivitamin/mineral supplement (Supradyn® Energy 3RDA) following a single intake and following daily intake for 4-weeks on subjective ratings of 'fatigue/stress', metabolism and blood biomarkers of cell damage following both exercise and demanding cognitive tasks, in healthy young male and female volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are physically active (i.e. exercise at least 2 times per week)
* Subjects are able to run non-stop on a treadmill at a moderate pace for 30mins
* Subjects agree to abstain throughout the trial from all dietary vitamin and mineral supplements
* Subjects are, in the opinion of the investigator, willing to participate in all scheduled visits and to adhere to all study procedures
* Subjects accept to refrain from alcohol intake 24 hours and to fast for a minimum of 10 hours before the study visits
* Subjects do not have a current diagnosis of a significant medical condition which may interfere with the subject's ability to perform assessments and successfully completes training
* Subjects provide a personally signed and dated informed consent indicating that the subject has been informed of all pertinent aspects of the trial and understood and accepts these
* Have a bank account (required for payment)

Exclusion Criteria:

* Smokers (smoking within the last 3 months)
* Blood pressure >140/90mmHg
* Excessive use of caffeine (> 500 mg caffeine per day) from all dietary sources
* Current intake of pharmaceuticals (excluding contraception)
* Have a recent history of (within 12 months of screening visit) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as more than 60g (men) / 40g (women) pure alcohol per day (7 / 5.5 units)
* A history of neurological or psychiatric diseases excluding anxiety or depression
* Current diagnosis of depression or anxiety
* A history of significant head trauma
* Have sleep disturbances and/or are taking sleep aid medication
* Have learning difficulties or dyslexia
* Have visual impairment that cannot be corrected with glasses or contact lenses
* Have frequent migraines that require medication (more than or equal to 1 per month)
* Have disorders of the blood (e.g. anemia, hemophilia, thrombocytosis)
* Have a heart disorder or a history of vascular illness
* Have a respiratory disorder that is induced by exercise or requires regular medication (Note: participants with asthma who only take their medication occasionally/as required are eligible for this study)
* Have type I or type II diabetes
* Have a history of renal or hepatic disease, or other severe diseases of the gastrointestinal tract (e.g. iron accumulation, iron utilization disorders, hypercalcaemia, hypercalciuria), that are likely to interfere with metabolism/absorption/secretion of the product under investigation
* Are pregnant, trying to get pregnant or breast feeding
* Have any health condition that would prevent fulfillment of the study requirements
* Any condition which may interfere with the subjects ability to perform assessments
* Are employed in a job that includes night shift work
* Participation in another clinical trial within 30 days prior to screening
* Have habitually supplemented with vitamins or minerals, within the last month (defined as more than 3 consecutive days or 4 days in total)
* BMI above 30 kg/m2
* Any history of hypersensitivity to the investigational product or its active or inactive constituents or any food allergy or intolerance

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Acute treatment effects on energy expenditure/metabolism during physical stress | Measures taken following acute treatment during exercise (45 minutes post acute treatment)
  ICa (Indirect Calorimetry) data obtained to determine energy expenditure, fat and carbohydrate oxidation
Acute treatment effects on energy expenditure/metabolism during mental stress | Measures taken following acute treatment during cognitive task performance (135 minutes post acute treatment)
  ICa (Indirect Calorimetry) data obtained to determine energy expenditure, fat and carbohydrate oxidation
Chronic treatment effects on energy expenditure/metabolism during physical stress | Measures taken following 28 days' chronic treatment, during exercise performance
  ICa (Indirect Calorimetry) data obtained to determine energy expenditure, fat and carbohydrate oxidation
Chronic treatment effects on energy expenditure/metabolism during mental stress | Measures taken following 28 days' chronic treatment, during cognitive task performance
  ICa (Indirect Calorimetry) data obtained to determine energy expenditure, fat and carbohydrate oxidation
Acute treatment effects on subjective arousal/stress/fatigue ratings as assessed by visual analogue scales during physical stress | Following acute treatment, measures taken before, after and every 10 minutes during 30 minute exercise period
  Subjective ratings of arousal (concentration, mental stamina/physical stamina) stress and fatigue (mentally tired/physically tired) visual analogue scales (scored along 100mm line)
Acute treatment effects on subjective arousal/stress/fatigue ratings as assessed by visual analogue scales during mental stress. | Following acute treatment, measures taken before, after and every 10 minutes during 30 minute cognitive task period
  Subjective ratings of arousal (concentration, mental stamina/physical stamina) stress and fatigue (mentally tired/physically tired) visual analogue scales (scored along 100mm line)
Chronic (28 days) treatment effects on subjective arousal/stress/fatigue ratings as assessed by visual analogue scales, during physical stress | Following 28 days' treatment, measures taken before, after and every 10 minutes during 30 minute exercise period
  Subjective ratings of arousal (concentration, mental stamina/physical stamina) stress and fatigue (mentally tired/physically tired) visual analogue scales (scored along 100mm line)
Chronic (28 days) treatment effects on subjective arousal/stress/fatigue ratings as assessed by visual analogue scales, during mental stress | Following 28 days treatment, measures taken before, after and every 10 minutes during 30 minute cognitive task period
  Subjective ratings of arousal (concentration, mental stamina/physical stamina) stress and fatigue (mentally tired/physically tired) visual analogue scales (scored along 100mm line)
Acute treatment effects on recovery biomarkers | Following acute treatment, taken at baseline and following exercise (75 minutes post-dose) and cognitive task performance (165 minutes post-dose). Then at 24h and 48hours post-exercise.
  Measuring levels of Interleukin-6, F2 isoprostanes, protein carbonyls, C-reactive protein, glutathione peroxidase, taken to assess recovery from exercise
Chronic (28 days) treatment effects on recovery biomarkers | Following 28 days treatment, taken at baseline, following exercise and cognitive task performance. Then at 24h and 48hours post-exercise.
  Measuring levels of Interleukin-6, F2 isoprostanes, protein carbonyls, C-reactive protein, glutathione peroxidase, taken to assess recovery from exercise

SECONDARY OUTCOMES:
Acute treatment effects on vitamin/mineral/homocysteine levels | Measured at baseline, then following acute treatment, after exercise (75 minutes post-dose)
  Measuring levels of Ferritin, vitamin B12, homocysteine, creatinine
Chronic (28 days) treatment effects on vitamin/mineral/homocysteine levels | Following chronic (28 days) treatment, measured after exercise
  Measuring levels of Ferritin, vitamin B12, homocysteine, creatinine
Acute treatment effects on cognitive performance | Following acute treatment, measured 135 minutes post dose
  Tasks include serial 3s, serial 7s and RVIP (Rapid Visual Information Processing), repeated 3 times
Chronic (28 days) treatment effects on cognitive performance | Following chronic (28 days) treatment
  Tasks include serial 3s, serial 7s and RVIP (Rapid Visual Information Processing), repeated 3 times

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Haskell-Ramsay, Dr, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne & Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dodd FL, Kennedy DO, Stevenson EJ, Veasey RC, Walker K, Reed S, Jackson PA, Haskell-Ramsay CF. Acute and chronic effects of multivitamin/mineral supplementation on objective and subjective energy measures. Nutr Metab (Lond). 2020 Feb 24;17:16. doi: 10.1186/s12986-020-00435-1. eCollection 2020. PMID 32123534